CLINICAL TRIAL: NCT01106456
Title: Culturally-Tailored Smoking Cessation for American Indians
Brief Title: Smoking Cessation for American Indians
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Won Choi, PhD, MPH (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Won Choi, PhD, MPH, Associate Professor, Preventive Medicine and Public Health, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11862; R01CA141618 (NIH)
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- All Nations Breath of Life (ANBL) (Experimental): All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT) then randomized into either the culturally-tailored "All Nations Breath of Life" program (ANBL) or Nontailored program (NT).
  Interventions: Behavioral: All Nations Breath of Life (ANBL); Drug: Pharmacotherapy
- Nontailored (NT) (Experimental): All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT) then randomized into either the culturally-tailored "All Nations Breath of Life" program (ANBL) or Nontailored program (NT).
  Interventions: Behavioral: Nontailored program (NT); Drug: Pharmacotherapy

INTERVENTIONS:
Behavioral: All Nations Breath of Life (ANBL) — ANBL consists of in-person group sessions and individual telephone calls. We have successfully conducted a pilot study of ANBL and have found very promising results. At six months and 12 months post baseline, all participants will be assessed for smoking status and smoking abstinence.
  Arms: All Nations Breath of Life (ANBL)
Behavioral: Nontailored program (NT) — The nontailored intervention includes the medicines listed above to all participants and targeted counseling delivered by non-American Indian counselors who have worked closely with the American Indian communities and respect the cultures, values, and traditions of the Indian people. Therefore, our intervention includes the current "best practice" recommendations for smoking cessation. At six months and 12 months post baseline, all participants will be assessed for smoking status and smoking abstinence.
  Other Names: Current best practices (CBP)
  Arms: Nontailored (NT)
Drug: Pharmacotherapy — All participants in the study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT)
  Other Names: Pharmacotherapy utilization

SUMMARY:
American Indians and Alaska Natives (AI/ANs) have the highest smoking rates of the major racial/ethnic groups in the United States, approaching 40% to 50%.1-3 In addition, this underserved population has very low smoking cessation and abstinence rates. The smoking-attributable mortality rate of AI/ANs is not only the highest but double that of other ethnic groups.4 To date, there have been almost no studies that have focused on methods to encourage smoking cessation among AI/AN smokers and no randomized clinical trials. There is a desperate need for effective, culturally tailored cessation programs.5, 6 We propose a 2 arm, group randomized clinical trial to be conducted at 2 sites in the Midwest (Kansas and Oklahoma).

We have begun to address these issues through the creation of the "All Nations Breath of Life" (ANBL) smoking cessation program using community-based participatory research methods. ANBL is group-based and is culturally-sensitive in all program components. It recognizes the sacred role of tobacco among many AI/ANs and how culture affects smoking cessation among AI/AN, while still addressing recreational smoking. Our pilot work shows promise for reducing cigarette smoking in AI/AN smokers, with quit rates of 30% at six months post-baseline, compared to 8-10% quit rates in other published studies.

All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline or Bupropion or NRT) then randomized into either the culturally-tailored "All Nations Breath of Life" program (ANBL) or Nontailored (NT. ANBL consists of in-person group sessions and individual telephone calls. We have successfully conducted a pilot study of ANBL and have found very promising results. At 6 months post baseline, all participants will be assessed for smoking status and continuous abstinence. We will randomize 28 groups per site (8 smokers per group) to ANBL or NT for a total sample size of 448 AI/AN smokers.

This study is the first controlled trial to examine the efficacy of a culturally-tailored smoking cessation program for AI/ANs. In collaboration with AI/AN colleagues in Oklahoma we designed and successfully piloted the intervention to be culturally-tailored and sustainable in order to enhance its potential for widespread adoption and ultimate impact among AI/AN smokers. If the intervention is successful, the potential health impact is significant because the prevalence of smoking is the highest in this population.

DETAILED DESCRIPTION:
This study will use a group randomized multi-site clinical trial design to examine the efficacy of a culturally-tailored smoking cessation program (ANBL) for AI/AN smokers versus Non-tailored (NT). AI/AN smokers in two sites (Kansas and Oklahoma) will be group randomized to either ANBL or Non-tailored (NT). Each site (KS and OK) will randomize 28 groups, resulting in 14 groups per arm of the intervention, per site. Participants in both groups (ANBL and NT) will be offered pharmacotherapy (e.g. varenicline or bupropion or NRT). The primary outcome of interest will be biochemically verified continuous abstinence at 1 year. Secondary endpoints include number of quit attempts and number of cigarettes smoked (among continuing smokers), pharmacotherapy utilization, and the number of completed group sessions. We will also examine the marginal cost-effectiveness of the intervention. The study will proceed in three phases over a five-year period. Phase I will consist of development and training. Phase 2 will be to conduct the randomized trial, and Phase 3 consists of data analysis and dissemination. Participants will be recruited from two sites: Kansas and Oklahoma. Although the ANBL arm is a group intervention and the NT arm is individual standard care, the unit of randomization will be at the group level (further discussed in the next section - Randomization process). Recruitment and randomization will be balanced by site: both sites will recruit until we reach our target sample size of 448 AI/AN smokers who are at least 18 years of age. Each site will randomize 28 groups (14 groups per arm) with 8 smokers in each group for a total site sample size of 224 smokers per site. Pharmacotherapy: The PI and site PI of this study along with our AI/AN community members agreed that all participants (ANBL and NT arms) had to be offered pharmacotherapy (varenicline or bupropion or NRT) as a component of the study design. This decision was a collaborative one between the AI/AN tribes and the investigators who have worked with this population. The AI/AN community will not accept placebo treatment, therefore, the interventions would not be acceptable or feasible to potential participants if a placebo was part of the study design. In addition, we believed it was ethically imperative that we provided smoking cessation interventions consistent with the current clinical practice guidelines for the treatment of tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have a home address and telephone number
* Willing to participate in all study components
* Willing to be followed for 6 months
* Smoked at least 100 cigarettes in their lifetime
* Current smoker
* American Indian or Alaska Native

Exclusion Criteria:

* Planning to leave the state within next 24 months
* Pregnant or breast feeding or planning to become pregnant in next 4 months.
* Medically ineligible after screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Choi, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Oklahoma College of Public Health, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi WS, Faseru B, Beebe LA, Greiner AK, Yeh HW, Shireman TI, Talawyma M, Cully L, Kaur B, Daley CM. Culturally-tailored smoking cessation for American Indians: study protocol for a randomized controlled trial. Trials. 2011 May 18;12:126. doi: 10.1186/1745-6215-12-126. PMID 21592347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Southern and Northern Plains regions, from reservations communities and in rural locations, including tribal trust land.
Pre-assignment Details: Exclusion criteria included intention to leave the state within the next 2 years, being pregnant/breastfeeding, planning to become pregnant in next 4 months, being medically ineligible after screening. Participants were recruited in April 2011, the final participant had their 6-month follow-up in July 2014.
Groups:
- All Nations Breath of Life Program (ANBL): All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT) then randomized into the culturally-tailored "All Nations Breath of Life" program (ANBL)
- Nontailored Program (NT): All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT) then randomized into the Nontailored program (NT).
Period: Overall Study
Arm/Group | All Nations Breath of Life Program (ANBL) | Nontailored Program (NT)
Started | 243 | 220
Completed | 140 | 96
Not Completed | 103 | 124

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | All Nations Breath of Life Program (ANBL) | Nontailored Program (NT) | Total
Number analyzed (Participants) | 243 | 220 | 463
Age, Categorical [Count of Participants; unit: Participants] — Population: The row populations only includes participants with available data.
  Participants
    number analyzed (Participants) | 226 | 215 | 441
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 212 | 206 | 418
    >=65 years | 14 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The row populations only includes participants with available data.
  years
    number analyzed (Participants) | 226 | 215 | 441
    (all) | 45.43 (12.98) | 43.12 (13.22) | 44.3 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The row populations only includes participants with available data.
  Participants
    number analyzed (Participants) | 230 | 217 | 447
    Female | 167 | 168 | 335
    Male | 63 | 49 | 112

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point Prevalence Abstinence From Smoking for 6 Months
Description: The primary outcome of the study was salivary cotinine-verified 7-day point prevalence smoking abstinence at 6 months (Have you smoked at least part of a cigarette in the past 7 days?) using responders-only analyses.
Time Frame: 6 months
Population: The difference in the "overall number of participants analyzed, "from the "number analyzed," in the ANBL arm, is due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | All Nations Breath of Life Program (ANBL) | Nontailored Program (NT)
Number analyzed (Participants) | 140 | 96
Participants
  Self-reported Responder Only: number analyzed (Participants) | 137 | 96
  Self-reported Responder Only | 49 | 26
  Cotinine verified Responder only: number analyzed (Participants) | 137 | 96
  Cotinine verified Responder only | 26 | 15

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the study (5 years).
Description: All-cause mortality cases were unrelated to the study medication of intervention components.
Groups:
- Experimental 1: All Nations Breath of Life Program (ANBL): All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT) then randomized into either the culturally-tailored "All Nations Breath of Life" program (ANBL) or Nontailored program (NT).
  Experimental 1: All Nations Breath of Life program (ANBL): ANBL consists of in-person group sessions and individual telephone calls. We have successfully conducted a pilot study of ANBL and have found very promising results. At six months and 12 months post baseline, all participants will be assessed for smoking status and smoking abstinence.
  Pharmacotherapy (e.g. Varenicline or Bupropion or NRT): Pharmacotherapy (e.g. Varenicline or Bupropion or NRT)
- Experimental 2: Nontailored Program (NT): All participants in the proposed study will be offered pharmacotherapy (e.g. Varenicline, Bupropion, or NRT) then randomized into either the culturally-tailored "All Nations Breath of Life" program (ANBL) or Nontailored program (NT).
  Experimental 2: Nontailored program (NT): The nontailored intervention includes the medicines listed above to all participants and targeted counseling delivered by non-American Indian counselors who have worked closely with the American Indian communities and respect the cultures, values, and traditions of the Indian people. Therefore, our intervention includes the current "best practice" recommendations for smoking cessation. At six months and 12 months post baseline, all participants will be assessed for smoking status and smoking abstinence.
  Pharmacotherapy (e.g. Varenicline or Bupropion or NRT): Pharmacotherapy (e.g. Varenicline or Bupropion or NRT)
Arm/Group | Experimental 1: All Nations Breath of Life Program (ANBL) | Experimental 2: Nontailored Program (NT)
All-Cause Mortality (participants affected / at risk) | 0/243 | 2/220
Serious Adverse Events (participants affected / at risk) | 0/243 | 0/220
Other Adverse Events (participants affected / at risk) | 7/243 | 8/220
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental 1: All Nations Breath of Life Program (ANBL) (N=243) | Experimental 2: Nontailored Program (NT) (N=220)
Sleep disturbance (General disorders) | 1 (1) | 2 (2) — Adverse event from participants taking varenicline.
Depression (General disorders) | 2 (2) | 2 (2) — Adverse event from participants taking varenicline.
Upset stomach (General disorders) | 1 (1) | 0 (0) — Adverse event from participants taking varenicline.
Nausea (General disorders) | 0 (0) | 1 (1) — Adverse event from participants taking varenicline.
Elevated blood pressure (General disorders) | 0 (0) | 1 (1) — Adverse event from participants taking varenicline.
Constipation (General disorders) | 1 (1) | 0 (0) — Adverse event from participants taking nicotine patch.
Aggressiveness and irritability (General disorders) | 1 (1) | 0 (0) — Adverse event from participants taking bupropion.
Skin reactions (General disorders) | 1 (1) | 0 (0) — Adverse event from participants taking bupropion and nicotine patch.
Chest pain (General disorders) | 0 (0) | 1 (1) — Adverse event from participants taking nicotine gum.
Chest pressure (General disorders) | 0 (0) | 1 (1) — Adverse event from participants taking nicotine patch.

LIMITATIONS AND CAVEATS:
Significant loss to follow-up, lower than expected salivary collection rates, lower long-term retention of participants, and higher than expected drop off from randomization to enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No